CLINICAL TRIAL: NCT03376399
Title: Do Sleeve Gastrectomies Result in Improved Gastric Emptying and Thus Improved Symptoms in Patients With Diabetic Gastroparesis?
Brief Title: Potential Benefits of Sleeve Gastrectomy Surgery on Diabetic Gastroparesis Symptoms
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled. Study terminated at PI's discretion
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 017-370
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Weight Loss; Diabetic Gastroparesis; Bariatric Surgery Candidate; Sleeve Gastrectomy; Gastric Emptying
Keywords: Sleeve Gastrectomy; Gastric Emptying; Diabetic Gastroparesis; Bariatric Surgery Candidate
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gastroparesis Cardinal Symptom Index Questionnaire — Patients with an established diagnosis of Diabetic Gastroparesis that are interested in a sleeve gastrectomy for weight loss will be asked to participate in the registry. Once the consent process is complete the patient will be asked to complete the Gastroparesis Cardinal Symptom Index Questionnaire prior to weight loss surgery and 30 days, 3 months, 6 months and 12 months after surgery.

SUMMARY:
The purpose of this registry is to evaluate if sleeve gastrectomy surgery will help with symptoms of delayed gastric emptying for patients suffering from diabetic gastroparesis.

DETAILED DESCRIPTION:
This is a prospective registry enrolling patients with an established diagnosis of diabetic gastroparesis and interested in receiving a sleeve gastrectomy for weight loss. An often intentional outcome of sleeve gastrectomy is an increase in gastric emptying. The relationship between how beneficial this outcome could be for diabetic gastroparesis patients suffering from delayed gastric emptying is not very well established. The purpose of this study is to find out if sleeve gastrectomy surgery will also help with symptoms of delayed gastric emptying. This study involves completing the Gastroparesis Cardinal Symptom Index questionnaire before your weight loss surgery and after surgery at the following time points; 30 days, 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* BMI > 35
* Diagnosis of diabetic gastroparesis as confirmed via scintigraphy
* Subject opting to undergo sleeve gastrectomy

Exclusion Criteria:

- Any previous weight loss surgery or prior gastrectomies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study group will be patients with diabetic gastroparesis who qualify for bariatric weight loss surgery (BMI >35, insurance/medicare bariatric coverage). These patients are referred by gastroenterologists and/or endocrinologists with established diagnosis of diabetic gastroparesis confirmed via delayed gastric emptying on scintigraphy. All available treatment options will be discussed with every qualifying patient. Patients opting for sleeve gastrectomy will be invited to participate in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Examine gastroparesis symptoms | 1 year
  Administer the Gastroparesis Cardinal Symptom Index (GCSI). The GCSI consists of three subscales: (1) Nausea/vomiting, (2) Fullness/early satiety, and (3) Bloating/distention. The average score is calculated from these three subscales with higher scores indicating greater symptom severity. The symptoms are rated on a scale from 0-5 with zero reflecting no symptoms and 5 indicating very severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Davis, DO, Principal Investigator — Baylor Scott & White, Baylor University Medical Center
Locations (1):
- Baylor Weight Loss Surgery Center, Dallas, Texas, United States